CLINICAL TRIAL: NCT00536172
Title: Prevention of Depression in Patients Being Treated for Head and Neck Cancer
Brief Title: Evaluating the Effectiveness of Escitalopram to Prevent Depression in Head and Neck Cancer Patients Receiving Treatment
Acronym: PROTECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0188-07-FB; R01MH079420 (NIH); DAHBR 96-BHC (Other Grant/Funding Number: National Institute of Mental Health (NIMH))
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Results first posted 2014-02-14 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Depression
Keywords: Antidepressant; Major depression; Prevention; Head and neck cancer
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Head and Neck Neoplasms | interventions — Escitalopram; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Experimental): Participants will receive treatment with escitalopram
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Participants will receive treatment with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — Participants take 10 mg for 1 week and then 20 mg for 15 weeks.
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Placebo — Placebo distribution matches the active medication.
  Other Names: Sugar pill; Inactive substance
  Arms: Placebo

SUMMARY:
This study will evaluate the effectiveness of escitalopram to prevent depression in head and neck cancer patients receiving treatment.

DETAILED DESCRIPTION:
Most types of head and neck cancer develop in the lining of cells found within many parts of the head and neck. Each year, more than 40,000 adults are diagnosed with head and neck cancer in the United States. The leading cause of this type of cancer is tobacco use. Common signs and symptoms of head and neck cancer include blood in saliva; frequent nose bleeds; and difficulty chewing, swallowing, or breathing. Effective treatments for head and neck cancer are available if the cancer is found in its early stages. However, treatment is difficult, causing many people to become depressed within 3 months of being diagnosed. Unfortunately, depression can lead to delays in treatment, impair quality of life, and decrease long-term survival. The purpose of this study is to determine whether the use of antidepressant medication initiated prior to starting treatment will prevent the onset of depression during treatment in non-depressed head and neck cancer patients. This study will also determine if escitalopram will maintain quality of life during treatment, improve participation in treatment, decrease delays and premature discontinuation of treatment, and reduce alcohol and tobacco use in patients with head and neck cancer.

All participants will attend an initial screening, followed by eight clinic visits. The first clinic visit will include completion of an interview and brief questionnaires regarding depression, mental and emotional health, alcohol and tobacco use, and quality of life. Participants will then be randomly assigned to receive 16 weeks of the antidepressant escitalopram or a placebo pill. Participants will take 10 mg of their assigned medication every day for the first week and then 20 mg of their assigned medication every day for the remaining 15 weeks. Participants will visit the clinic every 2 weeks during treatment, at which time they will answer questions similar to those asked at the initial visit. Any medication side effects will also be recorded at each visit. Once treatment has been completed, participants will visit the clinic three more times over a period of 12 weeks. Similar questions as those at treatment visits will be asked. Results from this study will be used to assess whether depression is preventable in head and neck cancer patients if antidepressant medication is initiated before treatment begins.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or recurrent epidermoid cancer of the head and neck
* Requires more than minimal therapy for treatment
* Able to read and write in English
* Willing to use an effective form of birth control throughout the study

Exclusion Criteria:

* Meets MINI criteria for major depression, schizophrenia, or bipolar illness or scores 24 or less
* Suicidal or psychotic
* Current allergy or hypersensitivity to citalopram or other SSRIs
* Treated with monoamine oxidase inhibitors 14 days prior to study entry
* Use of antidepressants within 1 week of study entry
* Pregnant or breastfeeding
* History of an adequate cancer operation, radiation, or chemotherapy within 6 months of study entry
* Diagnosed with melanoma or lymphoma cancer of the head and neck
* Currently participating in another research study involving a therapeutic intervention

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-12-01 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2012-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J Burke, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Result] Lydiatt WM, Bessette D, Schmid KK, Sayles H, Burke WJ. Prevention of depression with escitalopram in patients undergoing treatment for head and neck cancer: randomized, double-blind, placebo-controlled clinical trial. JAMA Otolaryngol Head Neck Surg. 2013 Jul;139(7):678-86. doi: 10.1001/jamaoto.2013.3371. PMID 23788218
- [Derived] Vita G, Compri B, Matcham F, Barbui C, Ostuzzi G. Antidepressants for the treatment of depression in people with cancer. Cochrane Database Syst Rev. 2023 Mar 31;3(3):CD011006. doi: 10.1002/14651858.CD011006.pub4. PMID 36999619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 298 patients were screened for possible study eligibility from January 6, 2008, to December 28, 2011. 160 subjects agreed to participate.
Pre-assignment Details: 12 of the 160 subjects who agreed to participate were not eligible: 9 QIDS or QIDS-C >/=11; 1 not able/willing to return for follow-up; 1 received antidepressants in the past week; 1 not diagnosed with epidermoid cancer and meets MINI criteria for depression. The remaining 148 subjects were randomized.
Period: Overall Study
Arm/Group | Escitalopram | Placebo
Started | 74 | 74
Completed | 60 | 65
Not Completed | 14 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Placebo | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (11.3) | 62.8 (12.5) | 63.0 (11.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 43 | 85
  >=65 years | 32 | 31 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 59 | 59 | 118
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 72 | 71 | 143
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 72 | 73 | 145
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 74 | 74 | 148
Clinical Stage [Number; unit: participants] — Clinical stage of cancer done using the AJCC manual on staging (2008 edition), based on TNM system. T stands for tumor (by size or extension into adjacent structures or subsites), N stands for nodal burden, M stands for distant metastasis (0 for none or 1 for any). Stage is assigned using all clinical material available to the surgeon at time of entry. Prognosis is dependent on stage and site of disease. Stage 1 was not allowed in the study due to very good prognosis and less treatment morbidity. Stage II is early stage disease. Late stage is III, IVA, IVB and IVC.
  participants
    II | 17 | 18 | 35
    III/IV | 57 | 56 | 113
Cancer Site [Number; unit: participants] — anatomical location of tumor
  participants
    oral | 29 | 36 | 65
    pharynx | 25 | 24 | 49
    skin | 9 | 8 | 17
    salivary gland | 6 | 5 | 11
    sinus | 5 | 1 | 6
Cancer Type [Number; unit: participants]
  squamous cell | 65 | 67 | 132
  salivary gland | 5 | 5 | 10
  skin | 4 | 0 | 4
  missing | 0 | 2 | 2
Initial Treatment Type (Surgery or Radiation) [Number; unit: participants]
  surgery, not biopsy | 42 | 39 | 81
  radiation with/without chemotherapy | 32 | 35 | 67

OUTCOME MEASURES:

1. Primary Outcome: Depression as Assessed by the Quick Inventory of Depressive Symptomatology-Self Rated 16 (QIDS-SR-16)
Description: Number of participants reaching pre-defined threshold on the QIDS-SR-16 of >/=11. The QIDS-SR-16 total score ranges from 0-27. Scores ranging from 0 to 10 correspond with no to mild depression, while scores >/= 11 correspond to moderate to severe depression.
Time Frame: Measured pre-treatment and at Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, and 28
Population: Evaluable subjects
Measure: Number; unit: participants
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 60 | 65
participants | 6 | 16

ADVERSE EVENTS:
Time Frame: 16 weeks of blinded and 12 weeks of open-label treatment
Arm/Group | Escitalopram | Placebo
All-Cause Mortality (participants affected / at risk) | 16/74 | 13/74
Serious Adverse Events (participants affected / at risk) | 16/74 | 13/74
Other Adverse Events (participants affected / at risk) | 47/74 | 49/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=74) | Placebo (N=74)
Nausea and vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (General disorders) | 4 (5) | 1 (1) — Secondary to diarrhea
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (1)
Fractured Leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dizziness/Syncope/Fall (General disorders) | 2 (2) | 2 (2)
GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mental Status Change (Nervous system disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Coronary Stenosis (Cardiac disorders) | 0 (0) | 1 (1)
G-tube Procedure Monitoring (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=74) | Placebo (N=74)
Diarrhea (Gastrointestinal disorders) | 6 | 4
Insomnia (General disorders) | 10 | 13
Mucositis (General disorders) | 9 | 14
Nausea and vomiting (General disorders) | 16 | 8
Rash (Skin and subcutaneous tissue disorders) | 1 | 7
Upper Respiratory Infection (Infections and infestations) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No